CLINICAL TRIAL: NCT00321594
Title: A Phase I/II Study of PXD101 in Patients With Unresectable Hepatocellular Carcinoma With Pharmacokinetic and Pharmacodynamic Evaluation
Brief Title: Belinostat in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00141; CTRG-HC06/21/05; N01CM62205 (NIH); CDR0000463519 (Registry Identifier: PDQ (Physician Data Query)); NCT01251445 (obsolete NCT alias)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: belinostat

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101

SUMMARY:
This phase I/II trial is studying the side effects and best dose of belinostat and to see how well it works in treating patients with liver cancer that cannot be removed by surgery. Belinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity (DLT) and establish the maximum tolerated dose (MTD) of PXD101 (belinostat) in patients with unresectable hepatocellular carcinoma (HCC). (Phase I) II. Assess the pharmacokinetic profiles of PXD101 in these patients. (Phase I) III. Assess tumor response in patients treated with this drug. (Phase II)

OUTLINE: This is a multicenter, dose-escalation phase I study followed by a phase II study.

PHASE I: Patients receive belinostat intravenously (IV) over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of belinostat until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive belinostat (as in phase I) at the MTD determined in phase I.

After completion of study therapy, patients are followed for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma that is not amenable to curative resection
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques OR as ≥ 10 mm with MRI or spiral CT scan
* No known brain metastases
* No clinical ascites or encephalopathy
* Life expectancy > 12 weeks
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.7 mg/dL
* Albumin ≥ 2.8 mg/dL
* ALT ≤ 5.0 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 6 times ULN
* Prothrombin time ≤ 4 sec above ULN
* Creatinine ≤ 1.6 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients use effective contraception
* No Child's-Pugh's grading Class C hepatic impairment
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to PXD101
* No marked baseline prolongation of QT/QTc interval, including the following:

  * Repeated demonstration of a QTc interval > 500 msec
  * Long QT Syndrome
* No ongoing or active infection
* No significant cardiovascular disease, including any of the following:

  * Unstable angina pectoris
  * Uncontrolled hypertension
  * Congestive heart failure related to primary cardiac disease
  * Condition requiring anti-arrhythmic therapy
  * Ischemic or severe valvular heart disease
  * Myocardial infarction within the past 6 months
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* At least 2 weeks since prior valproic acid
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent participation in another investigational study
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent use of any of the following:

  * Disopyramide
  * Dofetilide
  * Ibutilide
  * Procainamide
  * Quinidine
  * Sotalol
  * Bepridil
  * Amiodarone
  * Arsenic trioxide
  * Cisapride
  * Calcium channel blockers (e.g., lidoflazine)
  * Clarithromycin
  * Erythromycin
  * Halofantrine
  * Pentamidine
  * Sparfloxacin
  * Domperidone
  * Droperidol
  * Chlorpromazine
  * Haloperidol
  * Mesoridazine
  * Thioridazine
  * Pimozide
  * Methadone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2010-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, Principal Investigator — Chinese University of Hong Kong-Prince of Wales Hospital
Locations (2):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States
- Cancer Therapeutics Research Group, Singapore, Singapore

REFERENCES:
- [Derived] Yeo W, Chan SL, Mo FK, Chu CM, Hui JW, Tong JH, Chan AW, Koh J, Hui EP, Loong H, Lee K, Li L, Ma B, To KF, Yu SC. Phase I/II study of temsirolimus for patients with unresectable Hepatocellular Carcinoma (HCC)- a correlative study to explore potential biomarkers for response. BMC Cancer. 2015 May 12;15:395. doi: 10.1186/s12885-015-1334-6. PMID 25962426
- [Derived] Wang LZ, Ramirez J, Yeo W, Chan MY, Thuya WL, Lau JY, Wan SC, Wong AL, Zee YK, Lim R, Lee SC, Ho PC, Lee HS, Chan A, Ansher S, Ratain MJ, Goh BC. Glucuronidation by UGT1A1 is the dominant pathway of the metabolic disposition of belinostat in liver cancer patients. PLoS One. 2013;8(1):e54522. doi: 10.1371/journal.pone.0054522. Epub 2013 Jan 30. PMID 23382909

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Level 1: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose level: 600 mg/m2/day
- Phase I, Level 2: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose level: 900 mg/m2/day
- Phase I, Level 3: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose level: 1200 mg/m2/day
- Phase I, Level 4; Phase II, MTD Dose: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose level: 1400 mg/m2/day
Period: Phase I, Level 1-4
Arm/Group | Phase I, Level 1 | Phase I, Level 2 | Phase I, Level 3 | Phase I, Level 4 | Phase II, MTD Dose
Started | 3 | 3 | 6 | 6 | 0
Completed | 3 | 3 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase II, MTD Dose
Arm/Group | Phase I, Level 1 | Phase I, Level 2 | Phase I, Level 3 | Phase I, Level 4 | Phase II, MTD Dose
Started | 0 (Only last six patients in Phase I, Level 4 include in Phase II MTD Dose) | 0 (Only last six patients in Phase I, Level 4 include in Phase II MTD Dose) | 0 (Only last six patients in Phase I, Level 4 include in Phase II MTD Dose) | 6 (Only last six patients in Phase I, Level 4 include in Phase II MTD Dose) | 36 (last six patients in Phase I, Level 4 include in Phase II MTD Dose total number = 6 + 36 = 42)
Completed | 0 | 0 | 0 | 6 | 36
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 42 Patients from Phase II (including last 6 patients from Phase I)
Groups:
- Phase I: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV Level 1: Dose: 600mg/m2/day Level 2: Dose: 900mg/m2/day Level 3: Dose: 1200mg/m2/day
- Treatment (Enzyme Inhibitor Therapy): Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV Dose: 1400mg/m2/day
- Total: Total of all reporting groups
Arm/Group | Phase I | Treatment (Enzyme Inhibitor Therapy) | Total
Number analyzed (Participants) | 12 | 42 | 54
Age, Continuous [Median (Full Range); unit: year] | 54 [38 to 68] | 57.5 [35 to 76] | 56.5 [35 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 38 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 42 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 2 | 1 | 3
  United States | 0 | 1 | 1
  Hong Kong | 10 | 34 | 44
  South Korea | 0 | 5 | 5
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLT) and Maximum Tolerated Dose (MTD) of Belinostat in Patients With Inoperable HCC (Phase I)
Description: DLT is defined as any grade 4 hematological toxicity and any grade 3 or 4 non hematological toxicity during cycle 1, excluding alopecia. Specifically, grade 3 nausea, vomiting, or diarrhea that does not respond to therapy is considered dose-limiting. Also, delays in treatment greater than 2 weeks are also dose-limiting. MTD is defined as the dose below which >= 2 of 3 or >= 2 of 6 patients experience DLT. Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Course 1
Measure: Count of Participants; unit: Participants
Groups:
- Phase I, Level 1: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 600 mg/m2/day
- Phase I, Level 2: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 900 mg/m2/day
- Phase I, Level 3: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 1200mg/m2/day
- Phase I, Level 4: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 1400mg/m2/day
Arm/Group | Phase I, Level 1 | Phase I, Level 2 | Phase I, Level 3 | Phase I, Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Phase I, Level 1 vs Phase I, Level 2 vs Phase I, Level 3 vs Phase I, Level 4; MTD is defined as the dose below which >=2 of 3 or >= 2 of 6 patients experience DLT; Test type: Other; Maximum Tolerated Dose = 1400 — MTD was not reached and the maximum dose of 1400 mg/m2 is used in Phase II portion

2. Primary Outcome: Tumor Response in Patients With Inoperable HCC Using Belinostat (Phase II)
Description: Evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. The 95% confidence intervals should be provided.
Time Frame: Every 2 courses (approximately 6 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Phase II, MTD: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 1400mg/m2/day
Arm/Group | Phase II, MTD
Number analyzed (Participants) | 42
Participants
  Partial Response | 1
  Stable disease | 19
  Progressive disease | 22

ADVERSE EVENTS:
Time Frame: The adverse event data was assessed during treatment.
Description: the definition of adverse event and/or serious adverse event is same as clinicaltrials.gov definition The AE were only monitored for participants in Phase II portion.
Groups:
- Phase 1, Level 2: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 900mg/m2/day
- Phase I, Level 4: Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  belinostat: Given IV
  Dose: 600 to 1400mg/m2/day
Arm/Group | Phase I, Level 1 | Phase 1, Level 2 | Phase I, Level 3 | Phase I, Level 4 | Phase II, MTD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 1/42
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/42
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less